CLINICAL TRIAL: NCT04272775
Title: A Phase 1 Study of MLN9708 in Japanese Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of MLN9708 in Japanese Participants With Relapsed and/or Refractory Multiple Myeloma (RRMM)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision; No Safety Or Efficacy Concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TB-MC010034; JapicCTI-121822 (Registry Identifier: JapicCTI); U1111-1243-1737 (Registry Identifier: WHO)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Ixazomib 4.0 mg (Experimental): Ixazomib 4.0 milligram (mg), capsules, orally, once, on Days 1, 8, and 15 in 28-day treatment cycle for up to Cycle 87.
  Interventions: Drug: Ixazomib
- Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone (Experimental): Ixazomib 4.0 mg, capsules, orally, once, on Days 1, 8, and 15 in 28-day treatment cycle along with lenalidomide 25 milligram per day (mg/day), capsules, orally, once, from Days 1 to 21 and dexamethasone 40 mg/day, tablets, orally, once, on Days 1, 8, 15, and 22 in 28-day treatment cycle for up to Cycle 62.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort 3: Ixazomib 5.5 mg (Experimental): Ixazomib 5.5 mg, capsules, orally, once, on Days 1, 8, and 15 in 28-day treatment cycle for up to Cycle 87.
  Interventions: Drug: Ixazomib
- Cohort 4: Ixazomib 5.5 mg + Lenalidomide and Dexamethasone (Experimental): Ixazomib 5.5 mg, capsules, orally, once, on Days 1, 8, and 15 in 28-day treatment cycle along with lenalidomide 25 mg/day, capsules, orally, once, from Days 1 to 21 and dexamethasone 40 mg/day, tablets, orally, once, on Days 1, 8, 15, and 22 in 28-day treatment cycle for up to Cycle 87.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules.
  Other Names: MLN9708
Drug: Lenalidomide — Lenalidomide capsules.
  Arms: Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone; Cohort 4: Ixazomib 5.5 mg + Lenalidomide and Dexamethasone
Drug: Dexamethasone — Dexamethasone tablets.
  Arms: Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone; Cohort 4: Ixazomib 5.5 mg + Lenalidomide and Dexamethasone

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety, pharmacokinetics (PK) of ixazomib alone or in combination with lenalidomide and dexamethasone (Rd), and antitumor activity of ixazomib in participants with RRMM.

DETAILED DESCRIPTION:
The drug being tested in this study is called ixazomib. This study will evaluate the tolerability, safety, and PK of ixazomib administered alone or in combination with lenalidomide and dexamethasone in participants with relapsed and/or refractory multiple myeloma.

This study will enroll approximately 24 participants (3 to 6 participants in each dose-escalation cohort). Participants will be assigned to receive treatment in one of the four treatment cohorts:

* Cohort 1: Ixazomib 4.0 mg
* Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
* Cohort 3: Ixazomib 5.5 mg
* Cohort 4: Ixazomib 5.5 mg + Lenalidomide and Dexamethasone

This multi-center trial will be conducted in Japan. The overall time to participate in this study is approximately 7 years. Participants will make a final visit 29 days after receiving their last dose of drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese participants with multiple myeloma according to diagnostic criteria.
2. Previously treated with 2 or more regimens including all the following drugs; bortezomib, thalidomide or lenalidomide, corticosteroids.
3. Who have relapsed following the previous therapy or failed to continue the treatment due to their intolerability to the last treatment regimen for myeloma.
4. Measurable disease defined by at least one of the following 3 measurements; Serum M-protein: greater than or equal to (>=) 1 gram per deciliter (g/dL) (>= 10 gram per liter [g/L]), Urine M-protein: >= 200 mg/24 hours, Serum free light chain (FLC) assay: involved FLC level >= 10 milligram per deciliter (mg/dL) (>= 100 milligram per liter [mg/L]), provided that the serum FLC ratio is abnormal.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
6. 20 years or older at giving their informed consent.
7. Must be able to stay in the hospital for Cycle 1 treatment.
8. Must meet the following laboratory criteria at screening; Absolute neutrophil count (ANC): >=1,000 per cubic millimeter (/mm^3), Platelet count: >=75,000/mm^3, Total bilirubin: <=1.5* the upper limit of normal range (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST): less than or equal to (<=) 3* ULN, Creatinine clearance: calculated by using Cockcroft-Gault formula; MLN9708 monotherapy cohort: >=30 milliliter per minute (mL/min); MLN9708 with Rd cohort: >=60 mL/min.
9. Recovered (<= Grade 1) from the toxicities of the prior treatments. ANC >=1,000/mm^3.
10. Life expectancy of at least 3 months, in the judgment of the investigator.
11. Conforming to proper management guidelines of lenalidomide (MLN9708 with Rd cohort only).

Exclusion Criteria:

1. With plasmacytoma only.
2. With plasma cell leukemia.
3. With central nervous system invasion.
4. Radiotherapy within 14 days before enrollment.
5. Other anti-tumor drug administration within 21 days before enrollment.
6. Other investigational products administration within 21 days before enrollment (60 days from the last dose for carfilzomib).
7. Antibody treatment within 42 days before enrollment.
8. Systemic treatment with potent cytochrome P450 (CYP) isozyme 1A2 inhibitors (fluvoxamine, enoxacin), potent CYP3A inhibitors (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole), or potent CYP3A inducers (rifampin, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of foods containing Ginkgo biloba extract, St. John's Wort, or grapefruit within 14 days before enrollment.
9. Treatment with corticosteroids greater than (>) 10 mg of prednisolone per day. Inhaled and topical steroids are permitted.
10. Peripheral neuropathy >=Grade 2.
11. Diarrhea >= Grade 2.
12. Major surgery requiring general anesthesia within 14 days before enrollment.
13. Infection requiring systemic antibiotic treatment or other serious infections within 14 days before enrollment.
14. Evidence of concurrent uncontrolled cardiovascular conditions including hypertension, cardiac arrhythmias, New York Heart Association (NYHA) Class III or worse congestive heart failure, angina, myocardial infarction, or cerebral infarction within 6 months before enrollment.
15. Corrected QT interval (QTc) > 470 milliseconds on a 12-lead ECG obtained during the screening period.
16. Tested positive for human immunodeficiency virus (HIV) antibody, hepatitis B virus surface antigen (HBs antigen), or hepatitis C virus (HCV) antibody during the screening period.
17. Hypersensitivity to MLN9708 (including excipients), boron, or boron-containing drugs.
18. Hypersensitivity to lenalidomide, or dexamethasone, or excipients contained in the formulation of each drug (MLN9708 with Rd cohort only).
19. Known gastrointestinal diseases (difficulty swallowing, inflamed gastroenteritis, and Crohn disease), or gastrointestinal procedure (endoscopic procedure is permitted), that could interfere with the oral absorption or tolerance of the study treatment.
20. Uncontrolled diabetes mellitus.
21. A history of interstitial lung disease or lung fibrosis, or a current complication of interstitial lung disease or lung fibrosis diagnosed by diagnostic chest imaging.
22. Prior or current complications of deep vein thrombosis or pulmonary embolism (MLN9708 with Rd cohort only).

23 Diagnosed or treated for another malignancy within 2 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have complete resection.

24. Who do not consent to use adequate contraceptive precautions (example, condoms and oral contraceptives) during the following term:

* For women with childbearing potential, from when giving their consent through 3 months after the last dose of MLN9708, dexamethasone, or lenalidomide
* For men having their partners with childbearing potential, from giving their consent through 4 months after last dose of MLN9708, dexamethasone, or lenalidomide.

  25. Pregnant (example, positive for pregnancy test) or lactating. Lactation is prohibited from the first dose through 6 months after the last dose of MLN9708, dexamethasone, and lenalidomide.

  26. Use of an investigational medical device within 28 days before enrollment. 27. Any inabilities that could potentially interfere with the consent or completion of treatment according to this protocol.

  28. Having difficulties in participation to this study by the investigator's judgment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-06-05 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Japan from 05 June 2012 to 15 February 2019.
Pre-assignment Details: Relapsed and/or refractory multiple myeloma (RRMM) participants were enrolled to receive ixazomib 4.0 milligram (mg) in: Cohort 1 and along with lenalidomide 25 milligram per day (mg/day) and dexamethasone 40 mg/day (Rd) in Cohort 2. Study was terminated after completion of Cohorts 1 and 2 due to business decision; no safety or efficacy concerns.
Groups:
- Cohort 1: Ixazomib 4.0 mg: Ixazomib 4.0 mg, capsules, orally, once, on Days 1, 8, and 15 in 28-day treatment cycle for up to Cycle 87.
- Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone: Ixazomib 4.0 mg, capsules, orally, once, on Days 1, 8, and 15 in 28-day treatment cycle along with lenalidomide 25 mg/day, capsules, orally, once, from Days 1 to 21 and dexamethasone 40 mg/day, tablets, orally, once, on Days 1, 8, 15, and 22 in a 28-day treatment cycle for up to Cycle 62.
Period: Overall Study
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Started | 7 | 7
Completed | 0 | 0
Not Completed | 7 | 7
Not completed — Study Terminated by Sponsor | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Symptomatic Deterioration | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Progressive Disease | 3 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who received at least one dose of ixazomib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (4.20) | 60.3 (5.82) | 61.9 (5.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 7 | 7 | 14
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 156.49 (7.932) | 165.29 (8.245) | 160.89 (9.015)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 58.01 (8.477) | 58.01 (9.688) | 58.01 (8.745)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] | 1.585 (0.1438) | 1.628 (0.1652) | 1.607 (0.1504)
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors/researchers to assess how participant's disease is progressing, assess how disease affects daily living activities of participant and determine appropriate treatment and prognosis. 0=Actively able to do activities; 1=Restricted in physical activity, able to do light/sedentary work; 2=Ambulatory (greater than [>] 50 percent (%) of waking hours), capable of self care, unable to do any work activities; 3=Capable of limited self care, confined to bed >50% of waking hours; 4=Completely disabled, cannot do any self care, totally confined to bed; 5=dead.
  Participants
    0 | 6 | 6 | 12
    1 | 1 | 0 | 1
    2 | 0 | 1 | 1
Medical and Surgical History [Count of Participants; unit: Participants]
  Had history | 7 | 7 | 14
  No history | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLT:Any following adverse events (AEs) possibly related to ixazomib assessed by Common Terminology Criteria for AEs (CTCAE) version 4.03; Grade 4 neutropenia/thrombocytopenia lasting >7 consecutive days; Grade 3/greater neutropenia with fever/infections; Grade 3/greater thrombocytopenia with clinically significant bleeding; platelet count less than (<)10,000 per cubic meter(/mm^3); Grade 2 peripheral neuropathy with pain/Grade 3 or greater peripheral neuropathy; Grade 3/greater nonhematologic toxicities with exceptions of arthralgia/myalgia, fatigue lasting <7 days manageable nausea/emesis with antiemetic prophylaxis, diarrhea that is controlled with supportive care; treatment delay of >14 days at start of Cycle 2 due to failure of hematologic/nonhematologic recovery; Other Grade 2/greater ixazomib related nonhematologic toxicities required permanent discontinuation of ixazomib;Inability to receive at least 80% of planned lenalidomide doses due to the AEs related to ixazomib.
Time Frame: From Cycle 1 Day 1 until Cycle 2 Day 1 (Cycle length is equal to [=] 28 days)
Population: The DLT analysis set consisted of DLT evaluable participants who received at least one dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 6 | 6
Participants | 1 | 1

2. Primary Outcome: Number of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: Baseline up to 29 days after last dose of study drug (up to Cycle 87 Day 44) (Each Cycle length=28 days)
Population: The safety analysis set consisted of all participants who received at least one dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 7 | 7
Participants | 7 | 7

3. Primary Outcome: Number of Participants With Grade 3 or Higher TEAE Related to Body Weight
Description: Body weight abnormalities were graded using the CTCAE version 4.03. as: Grade 1 (Mild, asymptomatic or mild symptoms); Grade 2 (Moderate, minimal, local or noninvasive intervention indicated); Grade 3 (Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated); Grade 4 (Life-threatening consequences, urgent intervention indicated); Grade 5 (Death related to AE).
Time Frame: Baseline up to 29 days after last dose of study drug (up to Cycle 87 Day 44) (Each Cycle length=28 days)
Population: The safety analysis set consisted of all participants who received at least one dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Grade 3 or Higher TEAE Related to Vital Signs
Description: Vital signs were graded using the CTCAE version 4.03. as: Grade 1 (Mild, asymptomatic or mild symptoms); Grade 2 (Moderate, minimal, local or noninvasive intervention indicated); Grade 3 (Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated); Grade 4 (Life-threatening consequences, urgent intervention indicated); Grade 5 (Death related to AE).
Time Frame: Baseline up to 29 days after last dose of study drug (up to Cycle 87 Day 44) (Each Cycle length=28 days)
Population: The safety analysis set consisted of all participants who received at least one dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 7 | 7
Participants | 1 | 0

5. Primary Outcome: Number of Participants With Grade 3 or Higher TEAE Related to 12-lead Electrocardiograms (ECGs)
Description: 12-lead ECGs were graded using the CTCAE version 4.03. as: Grade 1 (Mild, asymptomatic or mild symptoms); Grade 2 (Moderate, minimal, local or noninvasive intervention indicated); Grade 3 (Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated); Grade 4 (Life-threatening consequences, urgent intervention indicated); Grade 5 (Death related to AE).
Time Frame: Baseline up to 29 days after last dose of study drug (up to Cycle 87 Day 44) (Each Cycle length=28 days)
Population: The safety analysis set consisted of all participants who received at least one dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Grade 3 or Higher Laboratory Tests Abnormalities
Description: Laboratory tests abnormalities were graded using the CTCAE version 4.03. as: Grade 1 (Mild, asymptomatic or mild symptoms); Grade 2 (Moderate, minimal, local or noninvasive intervention indicated); Grade 3 (Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated); Grade 4 (Life-threatening consequences, urgent intervention indicated); Grade 5 (Death related to AE).
Time Frame: Baseline up to 29 days after last dose of study drug (up to Cycle 87 Day 44) (Each Cycle length=28 days)
Population: The safety analysis set consisted of all participants who received at least one dose of ixazomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 7 | 7
Participants
  Grade 4: Neutrophils low | 0 | 2
  Grade 4: Leukocytes low | 0 | 1
  Grade 4: Lymphocytes low | 3 | 0
  Grade 4: Platelets low | 3 | 2
  Grade 4: Sodium low | 0 | 1
  Grade 4: Potassium low | 0 | 1
  Grade 3: Neutrophils low | 4 | 2
  Grade 3: Hemoglobin low | 2 | 2
  Grade 3: Leukocytes low | 3 | 2
  Grade 3: Lymphocytes low | 3 | 3
  Grade 3: Platelets low | 0 | 2
  Grade 3: Albumin low | 1 | 1
  Grade 3: Corrected calcium high | 0 | 1
  Grade 3: Sodium low | 1 | 0
  Grade 3: Potassium low | 1 | 0
  Grade 3: Phosphate low | 1 | 1

7. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Days 1 and 15 of Cycle 1: pre-dose and at multiple time points (15, 30, 60, and 90 minutes and 2, 4, 8, 24, 48, 96, and 168 hours) post-dose (Cycle length=28 days)
Population: The pharmacokinetic (PK) analysis set consisted of all participants who received at least one dose of ixazomib and has evaluable PK data. The PK analysis set where data at specified time points was available.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 7 | 7
nanogram per milliliter (ng/mL)
  Day 1 | 65.3 (54.6) | 32.9 (19.3)
  Day 15: number analyzed (Participants) | 5 | 6
  Day 15 | 68.8 (59.9) | 34.5 (42.0)

8. Secondary Outcome: Number of Participants Who Achieved Complete Response (CR), Very Good Partial Response (VGPR), and Partial Response (PR)
Description: Number of participants who achieved CR, PR, VGPR were assessed in accordance to International Myeloma Working Group Uniform Response Criteria for Multiple Myeloma. CR: No immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow. Normal serum free light chain (SFLC) ratio if disease measurable only by SFLC. VGPR: Serum and urine M-protein detectable by immunofixation but not electrophoresis or greater than or equal to (>=) 90% decrease in serum M-protein with urine M-protein <100 milligram per 24 hours (mg/24 hrs). If disease measurable only by SFLC, >= 90% decrease in the difference between involved and uninvolved FLC levels (dFLC). PR: >= 50% reduction of serum M-protein and >= 90% reduction in urine M-protein or to <200 mg/24 hrs, or a >= 50% decrease in dFLC. A >=50% decrease in the size of soft tissue plasmacytomas present at baseline
Time Frame: Baseline up to 29 days after last dose of study drug (up to Cycle 87 Day 44) (Each Cycle length=28 days)
Population: The response evaluable analysis set consisted of all participants who received at least one dose of ixazomib, have measurable disease at baseline, and at least one postbaseline response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 7 | 6
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: TEAEs are AEs that started after the first dose of study drug and no more than 29 days after the last dose of study drug (Cycle 87 Day 44)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1: Ixazomib 4.0 mg | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/7 | 2/7
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ixazomib 4.0 mg (N=7) | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone (N=7)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ixazomib 4.0 mg (N=7) | Cohort 2: Ixazomib 4.0 mg + Lenalidomide and Dexamethasone (N=7)
Neutropenia (Blood and lymphatic system disorders) | 6 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4
Leukopenia (Blood and lymphatic system disorders) | 5 | 4
Lymphopenia (Blood and lymphatic system disorders) | 6 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Vomiting (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Perianal erythema (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 1 | 1
Adenoviral conjunctivitis (Infections and infestations) | 0 | 1
Body tinea (Infections and infestations) | 0 | 1
Genital infection fungal (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urethritis (Infections and infestations) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Fatigue (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 1
Face oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
C-reactive protein increased (Investigations) | 2 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 2
Delirium (Psychiatric disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Phlebitis (Vascular disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Epidermolysis (Congenital, familial and genetic disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04272775/Prot_000.pdf
  • Statistical Analysis Plan (2014-02-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT04272775/SAP_001.pdf